CLINICAL TRIAL: NCT07255456
Title: Correlation Between Inferior Vena Cava Collapsibility Index and Serum Lactate in Poly-trauma Patients in Emergency Unite
Brief Title: Correlation Between Inferior Vena Cava Collapsibility Index and Serum Lactate in Poly-trauma Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Farid Esmael Haridy Mohamed (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Farid Esmael Haridy Mohamed, Resident doctor at Emergency Department Assiut University, Assiut University
Organization: Assiut University (Other)
Other Study IDs: IVC-CI & lactate in polytrauma
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Polytrauma Patients
Keywords: IVC-CI Lactate polytrauma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Abdominal ultrasound and Serum Lactate Level — Observational study there's no intervention
  Other Names: Abdominal ultrasound; ABG device

SUMMARY:
Polytrauma is defined as the presence of multiple traumatic injuries that may cause systemic physiological derangements and life-threatening conditions. Hypovolemia from blood loss is a major cause of death in polytrauma patients, and traditional methods of volume assessment like blood pressure and heart rate are frequently late indicators and may be deceptive due to compensatory mechanisms. Early identification of these causes is essential for prompt intervention.The non-invasive ultrasound-based Inferior Vena Cava Collapsibility Index (IVC-CI), which offers information on intravascular volume status, is one such tool. Variations in the IVC's width throughout the respiratory cycle are reflected in the IVC collapsibility index. A high degree of collapsibility in patients who are breathing on their own usually denotes low central venous pressure and potential hypovolemia. The use of IVC measures as a stand-in for preload evaluation and fluid responsiveness has been validated by numerous studies, particularly in emergency and critical care situations.

The primary sources of lactate, the conjugate base of lactic acid, are red blood cells and muscles during anaerobic metabolism (when oxygen is limited). It is created when the enzyme lactate dehydrogenase (LDH) transforms pyruvate, the byproduct of glycolysis, into lactate; Serum lactate is a known indicator of tissue hypoperfusion and anaerobic metabolism, and elevated lactate levels are commonly seen in individuals with repeated injuries due to tissue hypoxia. Higher rates of morbidity, mortality, and extended hospitalizations in intensive care have all been linked to trauma patients with elevated lactate levels [3,4].

Given that both IVC-CI and serum lactate levels are reflective of hemodynamic compromise, exploring a potential correlation between them in polytrauma patients is clinically relevant. If a reliable relationship is established, bedside ultrasound of the IVC could serve as a fast, real-time indicator of systemic hypoperfusion, offering a complementary or even alternative assessment when laboratory lactate measurements are delayed or unavailable.

Additionally, because point-of-care ultrasound (POCUS) is quick, non-invasive, and repeatable, its use in trauma procedures has been growing. Because of this, emergency physicians who want to make quick but well-informed judgments during the critical period of trauma care will find the IVC-CI especially appealing [6]. Finding relationships between biochemical indicators such as lactate and ultrasonographic results may offer a more thorough method of patient assessment, facilitating more effective triage and resuscitation techniques. The purpose of this study is to look at the relationship between serum lactate levels and the Inferior Vena Cava Collapsibility Index in patients with polytrauma who arrive at the emergency room. Developing this connection could help improve prognostication in this high-risk population and optimize early resuscitation procedures.

DETAILED DESCRIPTION:
Polytrauma is defined as the presence of multiple traumatic injuries that may cause systemic physiological. derangements and life-threatening conditions.

In US Polytrauma requiring major injury is estimated at around 54 cases per 1 million population per year and Overall in-hospital mortality among trauma discharges increased modestly from about 6.6% to 7.5% over the period of 1993-2012;in Egypt Trauma is estimated to account for ~8% of all deaths in Egypt, based on WHO estimates and national studies;in the Suez Canal University Hospital (Aug 2019-Mar 2020), trauma represented 5.3% of all emergency department cases, and among polytrauma cases: 44.4% were mild, 27.3% were life-threatening, Mortality was 56.0% for life-threatening cases and 6.9% for non-life-threatening polytrauma .In the Suez Canal University Hospital (Aug 2019-Mar 2020), trauma represented 5.3% of all emergency department cases, and among polytrauma cases 44.4% were mild, 27.3% were life-threatening ,mortality was 56.0% for life-threatening cases and 6.9% for non-life-threatening polytrauma . Assiut University, 2017 data): among 292 polytrauma patients, trauma-related mortality was around 20%.roughly half of deaths occurred early.

Hypovolemia from blood loss is a major cause of death in polytrauma patients, and traditional methods of volume assessment like blood pressure and heart rate are frequently late indicators and may be deceptive due to compensatory mechanisms. Early identification of these causes is essential for prompt intervention. As a result, there is increasing interest in using faster and more sensitive bedside instruments to direct resuscitation and track hemodynamic stability in trauma situations.

The non-invasive ultrasound-based Inferior Vena Cava Collapsibility Index (IVC-CI), which offers information on intravascular volume status, is one such tool. Variations in the IVC's width throughout the respiratory cycle are reflected in the IVC collapsibility index. A high degree of collapsibility in patients who are breathing on their own usually denotes low central venous pressure and potential hypovolemia. The use of IVC measures as a stand-in for preload evaluation and fluid responsiveness has been validated by numerous studies, particularly in emergency and critical care situations [1,2].

The primary sources of lactate, the conjugate base of lactic acid, are red blood cells and muscles during anaerobic metabolism (when oxygen is limited). It is created when the enzyme lactate dehydrogenase (LDH) transforms pyruvate, the byproduct of glycolysis, into lactate; Serum lactate is a known indicator of tissue hypoperfusion and anaerobic metabolism, and elevated lactate levels are commonly seen in individuals with repeated injuries due to tissue hypoxia. Higher rates of morbidity, mortality, and extended hospitalizations in intensive care have all been linked to trauma patients with elevated lactate levels [3,4].

Given that both IVC-CI and serum lactate levels are reflective of hemodynamic compromise, exploring a potential correlation between them in polytrauma patients is clinically relevant. If a reliable relationship is established, bedside ultrasound of the IVC could serve as a fast, real-time indicator of systemic hypoperfusion, offering a complementary or even alternative assessment when laboratory lactate measurements are delayed or unavailable.

Additionally, because point-of-care ultrasound (POCUS) is quick, non-invasive, and repeatable, its use in trauma procedures has been growing. Because of this, emergency physicians who want to make quick but well-informed judgments during the critical period of trauma care will find the IVC-CI especially appealing [6]. Finding relationships between biochemical indicators such as lactate and ultrasonographic results may offer a more thorough method of patient assessment, facilitating more effective triage and resuscitation techniques. The purpose of this study is to look at the relationship between serum lactate levels and the Inferior Vena Cava Collapsibility Index in patients with polytrauma who arrive at the emergency room. Developing this connection could help improve prognostication in this high-risk population and optimize early resuscitation procedures.

ELIGIBILITY:
Inclusion Criteria:

* ▪ Adult patients, both sex from 18 to 60 years old presented to the ED with blunt or penetrating polytrauma.

Polytrauma according ATLS defined as simultaneous injuries to at least two body systems, with at least one of the injuries being life-threatening or typically refers to patients with a high Injury Severity Score (ISS) of 16 or greater.

* Hemodynamically stable or unstable at the time of admission.
* Informed consent obtained from patient or next of kin.

Exclusion Criteria:

* ▪ Any polytrauma patient presented with cardiogenic or obstructive shock.

  * Patient is known to be cardiac that influence venous return.

    * Renal failure.
    * Chronic liver disease.
    * Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population will consist of adult patients (≥18 years) presenting to the emergency department with polytrauma. Patients must be hemodynamically stable enough to undergo bedside ultrasound assessment of the inferior vena cava.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Positive correlation between IVC-CI and serum lactate level | At presentation

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared."